CLINICAL TRIAL: NCT00932243
Title: Bacteremia in Intensive Care Unit (ICU) and the Role of Toll-Like-Receptors (TLRs)
Brief Title: Bacteremia in Intensive Care Unit (ICU)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Thessaly (Other)
Responsible Party: Zakynthinos E, Intensive Care Unit department University Hospital of Larisa
Other Study IDs: 845UT
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Bacteremia and Sepsis; Toll-Like-Receptors (TLRs)
Keywords: bacteremia; sepsis; Toll-Like-Receptors (TLRs)
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The presence of bacteremia and sepsis in percent of critically ill patients and none at all, associated with different expression and faction of Toll-Like-Receptors (TLRs.

DETAILED DESCRIPTION:
INTRODUCTION Bacteremia is associated with significant morbidity and mortality in critically ill patients and increased the length of hospitalization. Incidence of bacteremia in Intensive Care Units ranges from 8 to 10% and mortality 40%.

Risk factors for the development of bacteremia include the presence of central intravascular catheters, hemodialysis, the use of parenteral nutrition, urine catheters, endotracheal tubes, mechanical ventilation, underlying diseases like cancer, various immunocompromised states, mellitus diabetes, malnutrition, renal and liver failure, transplantations, surgery operations, burns.

The most common microbial pathogens which cause bacteremia are Gram negative pathogens, Pseudomonas species, Staphylococcus aureus, Klebsiella species, Pseudomonas aeruginosa, Candida albicans, Acinetobacter baumanii, Streptococcus pneumoniae.

Toll-like receptors (TLRs) are important for the activation of innate immunity against microbial pathogens. TLRs are transmembrane proteins and are composed of leukine rich extracellular domain, a short intramembrane segment and an intracytoplasmic domain. Intracytoplasmic domain is similar to that of interleukin-1 (IL-1) receptor.

In humans, they have been identified eleven types of recognizing specific pathogen-associated molecular patterns (PAMPs). TLR1 and TLR2 form a heterodimer recognizing bacterial tri-acylated lipopeptides of Gram-positive bacteria. TLR2 and TLR6 form another heterodimer recognizing di-acylated lipopeptides of Gram-positive bacteria. TLR4 is a heterodimer recognizing lipopolysacharedes (LPS)of Gram-negative bacteria while TLR5 is a receptor recognizing flagellae of Gram-negative bacteria. All these aforementioned types of TLRs are expressed on the outer surface of the cell membrane. TLR3, TLR7 TRL8 and TLR9 is a group of receptors expressed on an internal surface of the phagosomes formed in the cytoplasm after the ingestion of the pathogens.TLR3 recognizes viral dsRNA, TLR7 recognizes imidazol-quinollines, TLR8 recognize ssRNA and TLR9 recognize non-methylated bacterial CpG DNA. In addition to bacterial and viral CpG DNA, TLR9 is presumably involved in pathogenesis of autoimmune disorders. TLR10 and TLR11 are still under investigation, although TLR11 seem to recognize uropathogenic bacteria.

We suppose that the presence of bacteremia and sepsis in percent of critically ill patients and none at all, associated with different expression and faction of TLRs Searching of genetic polymorphisms of TLRs which associated with the presence of bacteremia and sepsis in ICU patients, probably will help us to clarify the pathophysiology of sepsis.

Aim

The study is a perspective cohort study which aimed to:

1. Search of genetic polymorphisms of TLRs which associated with the presence of bacteremia and sepsis in ICU patients
2. Estimate the incidence of bacteraemia
3. Search the microbiology of bacteremia
4. Correlate the incidence of bacteraemia with clinical parameter, significant for the nursing of critically ill patients in ICU like:

   Α) the duration of nursing Β) the outcome of nursing
5. Correlate the incidence of bacteraemia with probable risk factors like:

A) Bronchoscope B) Hemodialysis C) Mechanical ventilation D) Use of central intravascular catheters E) Tracheostomy F) Use of parenteral nutrition G) Use of central intravascular catheters with antiseptic substance

MATERIALS AND METHOD

Settings: The study will be performed in ICU, University Hospital of Larissa (10 beds).

Participants: Participants in the study will be all the patients who will be nursed in ICU for a two years period and they will be studied for all stay in ICU until their transfer to other ward or until their death. Criterion of exclusion of patients from the study will constitute the time of hospitalisation of patients that will be smaller than 24 hours.

Tools: The estimate of incidence of bacteremia but also the investigation of her microbiological explanation and the estimate of her repercussions for the patients it is used the Protocol of Bacteremia This protocol consist data as general elements, elements that concern the bacteremia as the samples, the micro-organisms, the resistance in the antibiotics, the mechanic ventilation, risk factors for growth of bacteremia, the empiric issuing of antibiotics but also the elements of outcomes of patients.

Diagnosis of bacteremia will be based on Centre of Disease Control end Prevention (CDC) criteria.

For the laboratorial detection of polymorphisms of TLR9 will be taken blood samples from the patients in the three first days of their nursing and will be sent in laboratory for analysis. For the laboratorial confirmation of bacteremia will be taken blood cultures or percutaneous or via intravenous catheters, which will be sent for analysis in the laboratory. Each result of blood culture will be also accompanied by the antibiogram according to which will be determined also the therapeutic form of antibiotics from the servant doctors. The reception of blood cultures will be realised in each change of central catheters and in the appearance of fever wave.

The follow-up of patients will become in daily base and essential information will be collected through the cards of nursing and the files of patients with the laboratorial results.

For the estimate of gravity of patients will be used APACHE II Score, Glasgow Scale, and SOFA Scale.

Statistic Analysis:

The statistic analysis of data will be realised with the use of computational parcel of SISS 15.0 for Windows. Data will be compared between bacteremia and no bacteremia groups. The investigation of relation of various potential risk factors with the repercussion of bacteremia, will be realised with the bivariate and multivariate analysis and the statistical method of simple accountant regression (simple Logistic Regression) and multiple accountant regression (multiple Logistic Regression). The odds ratio (OR) and linear coefficient will be calculated and presented with 95% CI. P<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* presence in Intensive Care Unit

Exclusion Criteria:

* Length of stay <24 hours

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will be nursed in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chatzi, RN,MSc,ICU, Principal Investigator — University Hospital Larisa
Locations (1):
- Zakynthinos E, Larissa, Mezourlo, Greece

REFERENCES:
- [Derived] Chatzi M, Papanikolaou J, Makris D, Papathanasiou I, Tsezou A, Karvouniaris M, Zakynthinos E. Toll-like receptor 2, 4 and 9 polymorphisms and their association with ICU-acquired infections in Central Greece. J Crit Care. 2018 Oct;47:1-8. doi: 10.1016/j.jcrc.2018.05.012. Epub 2018 May 25. PMID 29860039